CLINICAL TRIAL: NCT05747157
Title: Safety and Efficacy of Metabolically Armed CD19 CAR-T Cells (Meta10- 19) in the Treatment of r/r B-ALL Clinical Research
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: Leman Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Meta10-19-002
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-03

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: Meta10-19; CAR-T Cells Therapy; r/r B-ALL
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of Metabolically Armed CD19 CAR-T cells (Experimental): Patients undergo leukapheresis. Patients will receive a lymphodepletion chemotherapy with cyclophosphamide and fludarabine before CAR-T cells infusion. A dose of metabolically armed CD19 CAR-T cells will be infused on day 0.
  Interventions: Drug: Metabolically Armed CD19 CAR-T cells

INTERVENTIONS:
Drug: Metabolically Armed CD19 CAR-T cells — Each subject receive metabolically armed CD19 CAR-T cells by intravenous infusion.
  Other Names: Meta10-19

SUMMARY:
A Study of Metabolically Armed CD19 CAR-T Cells Therapy for Patients With Relapsed and/or Refractory B-cell Acute Lymphoblastic Leukemia

DETAILED DESCRIPTION:
This is a single arm , open-label study. This study is indicated for relapsed and/or refractory CD19+ B-cell Acute Lymphoblastic Leukemia . The selections of dose levels and the number of subjects are based on clinical trials of similar foreign products.

1. Main research objectives:

   To evaluate the safety and efficacy of metabolically armed CD19 CAR-T Cells in the treatment of r/r B-ALL.
2. Secondary research objectives:

A. To evaluate the pharmacokinetic (PK) and pharmacodynamics(PD) characteristics of metabolically armed CD19 CAR-T Cells after infusion.

B. To evaluate tumor remission after infusion of metabolically armed CD19 CAR-T Cells.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or his/her guardian voluntarily signed the informed consent；
2. Patients with relapsed and refractory B-cell Acute Lymphoblastic Leukemia.

   Definition of relapsed or refractory B-ALL (meeting one of the following conditions):
   1. 2 or more relapses;
   2. Bone marrow relapsed after allo-HSCT and prepared to infuse Meta10-19 more than 6 months after allo-HSCT ;
   3. CR not achieved after standardized chemotherapy;
   4. Philadelphia-chromosome-positive (Ph+) patients who are ineffective or intolerant to first- and second-generation tyrosine kinase inhibitor (TKI) treatments, or who have contraindications to tyrosine kinase inhibitors;
   5. The number of primordial cells (lymphoblast and prolymphocyte) in bone marrow is ≥ 5%
3. CD19 expression was positive by biopsy or flow cytometry (accept the results of this peripheral blood mononuclear cells collection or previous Class A tertiary hospital before this peripheral blood collection);
4. Expected survival time greater than 12 weeks
5. The baseline ECOG score was 0 or 1；
6. Organ function：

   1. Kidney function:

      Serum creatinine ≤1.5 times ULN, or； The glomerular filtration rate (eGFR) estimated by MDRD formula was ≥60m/min/1.73m2；[eGFR=186×（age）-0.203×SCr-1.154（mg/dl），for females, the result was ×0.742]；
   2. Liver function： ALT≤5 times ULN, and; Patients with total bilirubin ≤2.0mg/dl, except those with Gilbert-Meulengracht syndrome. Patients with Gilbert-.Meulengracht syndrome with total bilirubin ≤3.0 times ULN and direct bilirubin ≤1.5 times ULN were included.
   3. Pulmonary function: ≤CTCAE grade 1 dyspnea and oxygen saturation of blood (SaO2) ≥91% in indoor air environment.
7. Hemodynamic stability was determined by echocardiography or multichannel radionuclide angiography (MUGA) and LVEF ≥45％;
8. Patients using the following drugs must meet the following conditions:

   1. Steroid: Therapeutic doses of steroids must be discontinued 2 weeks prior to Meta10-19 infusion. However, physiological replacement doses of steroids are permitted, hydrocortisone or its equivalent < 6-12mg/mm2/ day；
   2. Immunosuppressive agent: Any immunosuppressive drug must be stopped ≥4 weeks before the informed consent is signed;
   3. Anti-proliferative therapy other than preconditioning chemotherapy is discontinued within 2 weeks prior to Meta10-19 infusion；
   4. Treatment for CNS disease must be stopped 1 week before Meta10-19 infusion (e.g., intrathecal methotrexate)
9. The patient has recovered from the toxicity of the previous treatment, that is, the CTCAE toxicity grade is less than 1 (The exception is specific toxicity of grade 2 or less, such as hair loss, which the researchers have determined is not recoverable in a short period of time) is suitable for pretreatment chemotherapy and CAR-T cell therapy;
10. Women of childbearing age and all male patients must consent to use an effective contraception for at least 12 months after Meta10-19 infusion and until two consecutive PCR tests show no more CAR-T cells in vivo.

Exclusion Criteria:

1. Patients with isolated extramedullary relapse;
2. Patients with confirmed diagnosis of Burkitt's lymphoma/ leukemia;
3. Patients who had received prophylaxis for CNS leukemia within 1 week prior to Meta10-19 infusion;
4. Patients with present or history of central nervous system diseases such as seizures disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement;
5. Patients with history of allogeneic hematopoietic stem cell transplantation (allo-HSCT) within 6 months prior to Meta10-19 infusion;
6. Patients who had received chemotherapy other than preconditioning chemotherapy within 2 weeks prior to Meta10-19 infusion ;
7. Patients who participated in other clinical trials within 30 days prior to enrollment;
8. Patients with active hepatitis B (defined as hepatitis B surface antigen positive or hepatitis B core antibody positive, concomitant hepatitis B virus DNA level > 1000 copies/ml) or hepatitis C (HCV RNA positive);
9. Patients with HIV antibody positive or treponema pallidum antibody positive;
10. Patients with uncontrolled acute life-threatening bacterial, viral or fungal infections (e.g. positive blood cultures ≤72 hours before Meta10-19 infusion)
11. Patients with unstable angina pectoris and/or myocardial infarction within 6 months prior to enrollment；
12. Patients with history of other malignancies, but the following conditions can be enrollment:

    1. Adequately treated basal or squamous cell carcinoma (requiring adequate wound healing before signing informed consent);
    2. Carcinoma in situ (DCIS) of cervical or breast cancer, which has been treated therapeutically, has shown no signs of recurrence for at least 3 years prior to the signing of the informed consent；
    3. The primary malignancy has been completely resected and in complete remission for ≥5 years。
13. Women who are pregnant or breastfeeding (pregnancy tests for women of childbearing age are positive);
14. Patients with active neuroautoimmune or inflammatory conditions (e.g. Guillian-Barre syndrome, amyotrophic lateral sclerosis);
15. Other conditions that the investigator considered should not be enrolled in this clinical study, such as poor compliance.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
MTD | MTD will be determined based on DLTs observed during the first 28 days of study treatment
  Determine the Maximal Tolerable Dose(MTD)
Objective response rate (ORR) | Within 3 months following infusion of Meta10- 19
  Measure Tumor response rate (including CR and PR)

SECONDARY OUTCOMES:
Pharmacokinetics | Up to 12 months after CAR-T treatment
  The number of CAR-T cells in peripheral blood was measured to evaluate the persistence of CAR-T cells
Pharmacodynamics | Up to 28 days after infusion
  Peak level of cytokines in peripheral blood

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu Q, Guo Y, Gao M, Xue L, Xu H, Li H, Zhang X, Liu C, Li Y, Chen Q, Ren J, Sathiyanadan K, Hu Y, Tang L, Huang H, Wang X. IL-10-expressing, anti-CD19 CAR T cells for patients with relapsed or refractory B-cell acute lymphoblastic leukaemia: an open-label, single-arm, phase 1 study. Lancet Haematol. 2025 Nov;12(11):e898-e907. doi: 10.1016/S2352-3026(25)00253-4. Epub 2025 Oct 16. PMID 41110448